CLINICAL TRIAL: NCT01478334
Title: Exercise-induced Improvements of Inflammatory Status in Patients With Rheumatoid Arthritis - Improvements of Cardiovascular Risk Factors and Quality of Life
Brief Title: Exercise-induced Improvements of Inflammatory Status in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RA-2011
Record Dates: First submitted 2011-09-07; First posted 2011-11-23 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Rheumatoid Arthritis
Keywords: High intensity exercise; cardiovascular risk factors
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise then control (Experimental)
  Interventions: Behavioral: high intensity interval training
- Control then exercise (Experimental)
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: high intensity interval training — First 10 week of high intensity interval training, twice a week. The interval training session consists of 10 minutes warm up at 70 percent of maximal heart rate and continues with 4 times 4 minutes of high intensity intervals at 90 to 95 percent of maximal heart rate separated by 3 minutes of active brakes in between at 70 percent of maximal heart rate. Training will be performed by cycling. Training intensity will be supervised through the use of polar puls monitors and the BORG scale of subjective perceived exhaustion.
  Second 10 weeks participants are instructed not to change their dietary patterns or physical activity levels during the study period.
  Arms: Exercise then control
Behavioral: Control — First 10 weeks participants are instructed not to change their dietary patterns or physical activity levels, and to continue their habitually lifestyle.
  Second 10 week of high intensity interval training, twice a week. The interval training session consists of 10 minutes warm up at 70 percent of maximal heart rate and continues with 4 times 4 minutes of high intensity intervals at 90 to 95 percent of maximal heart rate separated by 3 minutes of active brakes in between at 70 percent of maximal heart rate. Training will be performed by cycling. Training intensity will be supervised through the use of polar puls monitors and the BORG scale of subjective perceived exhaustion.
  Arms: Control then exercise

SUMMARY:
The primary aim of the study is to investigate if 10 weeks of high intensity interval training improve inflammatory status in patients with rheumatoid arthritis.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic, systemic inflammatory disorder that may affect many tissues and organs, but principally attacks synovial joints. Although the cause of rheumatoid arthritis is unknown, autoimmunity plays a role in both the chronicity and progression, and RA is considered as a systemic autoimmune disease.

Due to chronic inflammatory status, RA-patients are at higher risk of developing cardiovascular disease (CVD) compared to the general population. Accumulating evidence indicates that regular physical activity has beneficial effects on RA. The mechanisms behind exercise-induce improvements are none the less unclear and more research is needed to better understand the beneficial effects of exercise training in this patient group.

Recently, promising results from gene expression studies of blood cells have revealed unexplored fields of biomarker discovery and gene expression profiling of disease. Due to easy accessible and minimally invasive sample collection, gene expression profiling of whole blood might turn out to be a promising tool in molecular diagnostics and clinical medicine. To our knowledge, whole-genome transcriptional changes have not previously been studied in RA-patients undergoing a high-intensity exercise program.

Hypothesis: Ten weeks of high intensity interval training improves the inflammatory status, quality of life, and known risk factors for cardiovascular diseases.

In addition to measure traditionally inflammatory markers in the blood, whole genome analysis will be made.

ELIGIBILITY:
Inclusion Criteria:

* Ability to exercise
* written consent

Exclusion Criteria:

* Inability to exercise
* Known ischemic cardiovascular disease
* Severe pulmonary disease
* High activity level
* Pregnancy
* drug/alcohol abuse
* Unstable RA
* diagnosis before 2000

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2011-03; Primary Completion 2012-01 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Inflammatory markers in blood | 10 weeks
  C-reactive Protein (CRP), TNF-alfa, COMP, Pentraxin 3 using ELISA Whole-genome gene expression in blood cells using RNA(HumanHT-12 v4 Expression BeadChip)

SECONDARY OUTCOMES:
Endothelial function | 10 weeks
  Flow mediated dilatation (FMD).
quality of life | 10 weeks
  Questionnaire SF-36
HDL | 10 weeks
  Standard biochemical analysis procedure at St.Olavs hospital
Total Cholesterol | 10 weeks
  Standard biochemical analysis procedure at St.Olavs hospital
Blood glucose | 10 weeks
  Standard biochemical analysis procedure at St.Olavs hospital
whole-genome gene expression in blood cells | 10 weeks
  total RNA isolated from whole blood (Qiagen, Bioanalyzer, NanoDrop). Gene expression analysis on HumanHT-12 v4 Expression BeadChip.

CONTACTS AND LOCATIONS:
Overall Officials: Dorthe Stensvold, Study Director
Locations (1):
- Norwegian University of Science and Technology, Faculty of medicine, Department of circulation and medical imaging,, Trondheim, Norway

REFERENCES:
- [Result] Sandstad J, Stensvold D, Hoff M, Nes BM, Arbo I, Bye A. The effects of high intensity interval training in women with rheumatic disease: a pilot study. Eur J Appl Physiol. 2015 Oct;115(10):2081-9. doi: 10.1007/s00421-015-3186-9. Epub 2015 May 27. PMID 26013051